CLINICAL TRIAL: NCT03486288
Title: Kognitive Störungen Nach Elektiver Wirbelsäulenchirurgie Bei Älteren
Brief Title: Cognitive Impairment Following Elective Spine Surgery
Acronym: CONFESS
Status: Terminated | Type: Observational
Why Stopped: Recruitment delayed because of Sars-CoV-2 pandemic, elective surgery stopped, funding for undefinite extension not available
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB 192/17
Record Dates: First submitted 2018-03-01; First posted 2018-04-03 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Cognitive Impairment; Postoperative Delirium; Spine Fusion
Keywords: delirium; postoperative cognitive dysfunction; spine surgery; elderly; neuroinflammation; magnetic resonance imaging; resting state fmri; cerebral vasculature; quality of life
MeSH Terms: conditions — Cognitive Dysfunction; Emergence Delirium; Delirium; Postoperative Cognitive Complications; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium
- No Delirium

SUMMARY:
Older people are a rapidly growing proportion of the world's population and their number is expected to increase twofold by 2050. When these people become patients that require surgery, they are at particular high risk for postoperative delirium (POD), which is associated with longer hospital stays, higher costs, risk for delayed complications and cognitive dysfunction (POCD). Having suffered an episode of delirium is furthermore a predictor of long-term care dependency. Despite these risks, an increasing number of elderly undergo major elective surgery. This is reflected by the frequency of elective spinal surgery, in general, and instrumented fusions, in particular, which has markedly increased over the past few decades.

It is yet insufficiently understood, which, particularly modifiable, factors contribute to the development of POD and POCD following these major but plannable surgeries. A better understanding of risk factors would facilitate informed patient decisions and surgical strategies could be tailored to individual risk profiles.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years
* scheduled for elective spine surgery without opening the dura
* patient can give informed consent him-/herself
* German native speaker

Exclusion Criteria:

* dementia or neurodegenerative disease
* psychiatric disease
* prescription of CNS-active medication (e.g. antidepressants, antipsychotics, sedatives, alpha-1-antagonists)
* impossible to participate in follow-up
* participation in an interventional trial
* electronic or displacable metallic implants
* active neoplasm

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients seen in a neurosurgical oupatient clinic will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
postoperative delirium - incidence | ≤ 3 days postoperatively
  screening through Nu-DESC (Nursing Delirium Screening Scale) ≥ 2 and verification of screening procedure by DSM-V (Diagnostic and Statistical Manual of Mental Disorders 5th Edition) criteria once during each shift

SECONDARY OUTCOMES:
postoperative delirium - duration | ≤ 3 days postoperatively or until delirium resolves
  screening through Nu-DESC ≥ 2 and verification of screening procedure by DSM-V criteria DSM-V once during each shift
postoperative delirium - severity | ≤ 3 days postoperatively or until delirium resolves
  rated through CAM-S (Confusion Assessment Method - Severity) if patient was identified to be delirious
postoperative cognitive dysfunction - severity | baseline and 3 months postoperatively
  CERAD-Plus (Consortium to Establish a Registry for Alzheimer's Disease - Plus)
pre- and postoperative intelligence | baseline and 3 months postoperatively
  MWT-B (Mehrfachwahl-Wortschatz-Intelligenztest - B)
Markers of systemic inflammation | ≤ 2 days postoperatively
  C-reactive protein, Interleukins, Tumor necrosis factor among others
Markers of neuroinflammation | ≤ 2 days postoperatively
  Glial fibrillary acidic protein among others
Markers of oxidative and metabolic stress | ≤ 2 days postoperatively
  Malondialdehyd
Patient Reported Quality of life | baseline and 3 months postoperatively
  PROMIS-29 (Patient-Reported Outcomes Measurement Information System- Profile 29 incl. proxy-rating)
Patient Reported Quality of life - 2 | baseline and 3 months postoperatively
  SF-36 (Short Form 36)
Anxiety and depression | baseline and 3 months postoperatively
  HADS (Hospital Anxiety and Depression Scale)
Frailty | baseline and 3 months postoperatively
  Groningen Frailty Scale
Structural magnetic resonance imaging | baseline and 3 months postoperatively
  White matter lesions
Functional magnetic resonance imaging | baseline and 3 months postoperatively
  Resting state networks
Cerebral vasculature | baseline
  Ultrasound of extra- and intracranial cerebral arteries
Genetic polymorphisms | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fleischmann, MD, Principal Investigator — Department of Neurology; Jonas Müller, MD, Principal Investigator — Department of Neurosurgery
Locations (1):
- Department of Neurology, Greifswald, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Derived] Muller J, Nowak S, Vogelgesang A, von Sarnowski B, Rathmann E, Schmidt S, Rehberg S, Usichenko T, Kertscho H, Hahnenkamp K, Floel A, Schroeder HW, Muller JU, Fleischmann R. Evaluating Mechanisms of Postoperative Delirium and Cognitive Dysfunction Following Elective Spine Surgery in Elderly Patients (CONFESS): Protocol for a Prospective Observational Trial. JMIR Res Protoc. 2020 Feb 13;9(2):e15488. doi: 10.2196/15488. PMID 32053113